CLINICAL TRIAL: NCT05514990
Title: A Phase 1b/2 Study of Standard Doses of Bortezomib and Pembrolizumab ± Reovirus (Pelareorep) Combination Therapy in Patients With Relapsed Multiple Myeloma (AMBUSH Study)
Brief Title: Bortezomib and Pembrolizumab With or Without Pelareorep for the Treatment of Relapsed or Refractory Multiple Myeloma, AMBUSH Trial
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16M-22-1; NCI-2022-06505 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16M-22-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2022-08-19; First posted 2022-08-25 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; reolysin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (standard therapy) (Experimental): Patients receive bortezomib SC) or IV and dexamethasone PO, IV, or IM on days 1, 8, and 15 of each cycle. Patients also receive pembrolizumab IV over 30 minutes on day 9 of each cycle. Treatment repeats every 21 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Biological: Pembrolizumab
- Cohort II (standard therapy, pelareorep) (Experimental): Patients receive bortezomib SC or IV and dexamethasone either PO, IV, or IM on days 1, 8, and 15 of each cycle. Patients also receive pelareorep IV over 60 minutes on days 1, 2, 8, 9, 15, and 16 and pembrolizumab IV over 30 minutes on day 9 of each cycle. Treatment repeats every 21 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Biological: Pelareorep; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Bortezomib — Given SC or IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Dexamethasone — Given PO, IV, or IM
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Biological: Pelareorep — Given IV
  Other Names: PO BB0209; PO-BB0209; Reolysin; Reovirus Serotype 3; Wild-type Reovirus
  Arms: Cohort II (standard therapy, pelareorep)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I/II trial studies the safety of the combination of bortezomib, dexamethasone, and pembrolizumab with or without pelareorep in treating patients with multiple myeloma that has come back (relapsed) or does not response to treatment (refractory). Chemotherapy drugs, such as bortezomib and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. A virus modified in the laboratory, such as pelareorep, may be able to kill cancer cells without damaging normal cells. Giving the combination of bortezomib, dexamethasone, and pembrolizumab with pelareorep may work better in treating patient with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the safety of bortezomib-dexamethasone (BOR-D) and pembrolizumab (cohort 1) and its combination with pelareorep (PELA) (cohorts 2). (Phase 1B) II. To determine the recommended phase 2 dose (RP2D) for PELA in combination with BOR-D and pembrolizumab in patients with relapsed or refractory multiple myeloma (RRMM; cohorts 2). (Phase 1B) III. To estimate the efficacy of the combination of PELA, BOR -D and pembrolizumab in patients with RRMM. (Phase 2)

SECONDARY OBJECTIVES:

I. To evaluate the efficacy PELA in combination with BOR-D and pembrolizumab (cohorts 2) in patients with RRMM. (Phase 1B) II. To characterize the safety and tolerability of the combination, including acute and chronic toxicities. (Phase 2)

EXPLORATORY OBJECTIVES:

I. To compare changes in the tumor microenvironment (TME) and immune responses in patients treated with BOR-D and pembrolizumab (cohort 1) to patients treated with PELA, BOR-D, and pembrolizumab (cohort 2). (Phase 1B) II. To evaluate changes in the TME and immune responses in patients treated with the combination of PELA, BOR-D and pembrolizumab. (Phase 2)

OUTLINE: This is a phase IB dose escalation study followed by a phase II study. Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients receive bortezomib subcutaneously (SC) or intravenously (IV) and dexamethasone orally (PO), IV, or intramuscularly (IM) on days 1, 8, and 15 of each cycle. Patients also receive pembrolizumab IV over 30 minutes on day 9 of each cycle. Treatment repeats every 21 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients receive bortezomib SC or IV and dexamethasone either PO, IV, or IM on days 1, 8, and 15 of each cycle. Patients also receive pelareorep IV over 60 minutes on days 1, 2, 8, 9, 15, and 16 and pembrolizumab IV over 30 minutes on day 9 of each cycle. Treatment repeats every 21 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study, patients are followed-up every 12 weeks or every 6 months depending on status of disease.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory multiple myeloma (MM) after at least 3 previous lines of therapy. Previous treatment must have included a proteasome inhibitor (bortezomib, ixazomib or carfilzomib), an immunomodulatory agent (thalidomide, lenalidomide or pomalidomide) and an anti cd38 monoclonal antibody.
* Histologically confirmed diagnosis of MM with measurable disease, as defined by the presence of monoclonal immunoglobulin protein in serum electrophoreses of at least 0.5 g/dL for immunoglobulin G (IgG) or 0.25 g/dL for IgA, or measurable light chain in serum (100 mg/L) or urinary excretion of at least 200 mg monoclonal light chain per 24 hours.
* No continuing acute toxic effects (except alopecia) of any prior chemotherapy, radiotherapy or surgical procedures. All such effects must have resolved to Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 grade =< 1. Surgery (except minor procedures such as biopsies, intravenous [IV]-line placement, etc.) must have occurred at least 28 days prior to study enrollment.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
* Male or female >= 18 years of age at the time of signing the informed consent form (ICF).
* Life expectancy of at least 3 months.
* Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of relapse, refractory multiple myeloma will be enrolled in this study.
* A male participant must agree to use a contraception during the treatment period and for at least 7 months after the last dose of study treatment and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 7 months after the last dose of study treatment.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial, indicating that the patient is aware of the neoplastic nature of their disease and have been informed of the procedures of the protocol, the experimental nature of the therapy, possible alternative therapies, potential benefits, side effects, risks, and discomforts.
* Be willing and able to comply with scheduled visits, the treatment plan, and laboratory tests.
* Absolute neutrophil count (ANC) >= 1000/uL (collected within 10 days prior to the start of study intervention).
* Platelets >= 50,000/uL (collected within 10 days prior to the start of study intervention).
* Hemoglobin >= 8.0 g/dL or >= 5.0 mmol/L.
* Creatinine =< 1.5 x upper limit of normal (ULN) or measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance ([CrCl]) >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN (collected within 10 days prior to the start of study intervention).
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (collected within 10 days prior to the start of study intervention).
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase) [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase) [SGPT]) =< 2.5 x ULN (=< 5 x ULN for participants with liver metastases) (collected within 10 days prior to the start of study intervention).
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants (collected within 10 days prior to the start of study intervention).
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (collected within 10 days prior to the start of study intervention).
* Proteinuria normal or grade 1 based on 24-urine collection test. Patients with proteinuria >= grade 2 due to light chains in the urine may be eligible based on review of screening urine electrophoresis results.
* Thyroid-stimulating hormone (TSH), thyroxine (T4) and adrenocorticotropic hormone (ACTH) within normal limits. Patients under treatment for hormonal abnormality(s) will be individually assessed for inclusion based on their history and current status.
* Criteria for known Hepatitis B and C positive subjects. Hepatitis B and C screening tests are not required unless:

  * Known history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
  * As mandated by local health authority.
* Hepatitis B positive subjects:

  * Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.
  * Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.
* Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.

  * Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization.

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

  * Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.

  * Note: Participants must have recovered from all AEs due to previous therapies to =< grade 1 or baseline. Participants with =< grade 2 neuropathy may be eligible. Participants with endocrine -related AEs grade =< 2 requiring treatment or hormone replacement may be eligible.
  * Note: If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-central nervous system (CNS) disease. Palliative radiotherapy is allowed while on study treatment for treatment of symptomatic lesions.
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, bacillus calmette-guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.

  * Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Known additional malignancy that is progressing or has required active treatment within the past 5 years.

  * Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) or other noninvasive or indolent hat have undergone potentially curative therapy are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV) infection.

  * Note: No HIV testing is required unless mandated by local health authority.
* Concurrent active hepatitis B (defined as HBsAg positive and/or detectable HBV deoxyribonucleic acid [DNA]) and hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV ribonucleic acid [RNA]) infection.

  * Note: Hepatitis B and C screening tests are not required unless:

    * Known history of HBV and HCV infection.
    * As mandated by local health authority.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.
* History or prior allogenic stem cell transplant.
* Receipt of concurrent immunosuppressive therapy.
* Clinically significant cardiac disease (New York Heart Association, Class III or IV) including pre-existing arrhythmia, uncontrolled angina pectoris, myocardial infarction 1 year prior to study entry, or a known history of grade 2 or higher compromised left ventricular ejection fraction.
* Dementia or altered mental status that would prohibit informed consent.
* Has a history of or current evidence of any other severe, acute or chronic medical or psychiatric condition, therapy or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the principal investigator, would make the patient inappropriate for this study.
* History of allergic (anaphylactic) sensitivity to bortezomib, boron or mannitol.
* Grade 2 or greater neuropathy at the time of screening.
* Has a known history of active TB (Bacillus tuberculosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2026-08-22 (Estimated); Study Completion 2027-08-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) (Phase 1B) | During the 21 days of cycle 1
  Incidence of dose-limiting toxicities resulting from pelareorep (PELA) in combination with bortezomib-dexamethasone (BOR-D) and pembrolizumab will be assessed. Severity of Adverse Events (AEs) will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Incidence and severity of adverse events (AEs) (Phase 1B) | Up to 30 days following cessation of study intervention
  Incidence and severity of adverse events (AEs) will be graded according to NCI CTCAE version 5.0, and changes in clinical laboratory parameters.
Overall response rate (ORR) (complete response [CR] + partial response [PR]) (Phase 2) | Up to 3 years
  Overall response rate, complete response partial response per the International Myeloma Working Group (IMWG) Uniform Response Criteria for multiple myeloma (MM).

SECONDARY OUTCOMES:
ORR (CR + PR) (Phase 1B) | Up to 3 years
  ORR (CR + PR) per the IMWG Uniform Response Criteria for MM
Duration of response (DOR) (Phase 2) | Up to 3 years
  Time from first documentation of response (PR or greater) to first documentation of progressive disease (PD) or death from any cause, whichever occurs first.
Progression-free survival (PFS) (Phase 2) | Up to 3 years
  Time from the date of first study treatment to the date of first documented Progressive Disease (PD), as defined in the International Myeloma Working Group (IMWG) criteria, or death due to any cause, whichever occurs first.
Overall survival (OS) (Phase 2) | Up to 3 years
  Defined as the time from the first study treatment administration to death from any cause.
Incidence of adverse events (Phase 2) | From the time of intervention allocation through 90 days following cessation of study intervention or 30 days following cessation of study intervention
  Type, frequency, and severity of AEs, using the NCI CTCAE version 5.0.
Severity of serious adverse events (Phase 2) | From the time of intervention allocation through 90 days following cessation of study intervention or 30 days following cessation of study intervention
  Serious adverse events (SAEs), using the NCI CTCAE version 5.0.

OTHER OUTCOMES:
Changes in gene expression (Phase 1B, Phase 2) | Up to 3 years
  Will identify biological changes between pre-treatment and on-treatment biopsies as defined by changes in gene expression within the tumor microenvironment (TME).
Changes in the T cell repertoire within peripheral blood and the TME (Phase 1B, Phase 2) | Up to 3 years
  Will compare changes in the T cell repertoire within peripheral blood and the TME between pre-treatment and on-treatment biopsies, examining the formation of novel clones and the expansion of existing clones.
Changes in the expression of immune-related biomarkers (Phase 1B, Phase 2) | Up to 3 years
  To examine changes in the expression of immune-related biomarkers between pre-treatment and on-treatment blood samples and biopsies such as changes in programmed death protein-1 (PD-1) and programmed death ligand-1 (PDL-1) expression by immunohistochemistry (IHC) and imaging mass cytometry.
PELA in combination with different therapies (Phase 1B, Phase 2) | Up to 3 years
  Will evaluate whether PELA in combination with different therapies induces changes in different immune blood markers between pre-treatment and on-treatment blood samples (e.g., peripheral blood mononuclear cells [PBMCs]-flow cytometry and flow mass cytometry).
CD4 and CD8 T-cell reactivity (Phase 1B, Phase 2) | Up to 3 years
  Will examine CD4 and CD8 T-cell reactivity toward antigens and other stimuli between pre-treatment and on-treatment bone marrow biopsies and peripheral blood.
Number of effector T-cells and resting T-cells (Phase 1B, Phase 2) | Up to 3 years
  Will evaluate the number of effector (interferon-gamma [IFN-gamma] and Granzyme B) T-cells and resting T-cells in pre-treatment and on-treatment bone marrow biopsies and peripheral blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Kelly, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California